CLINICAL TRIAL: NCT03467464
Title: The Efficacy of EMDR in Youngsters With Autism: an Explorative Study
Brief Title: The Efficacy of EMDR in Youngsters With Autism
Acronym: EYE-catcher
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karakter Kinder- en Jeugdpsychiatrie (Other)
Collaborators: Fonds Psychische Gezondheid (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL6002609116
Record Dates: First submitted 2017-10-06; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2017-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism, EMDR; Children
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): EMDR treatment
  Interventions: Other: Eye Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Other: Eye Movement Desensitization and Reprocessing (EMDR) — The intervention consists of 10 weekly EMDR sessions of 60 minutes and targets stressful daily life (i.e. a situation that caused anger, fear or confusion) events rather than traumatic images from the past. For each session, a standardised EMDR protocol is used that consists of the following consecutive steps: 1) determining and visualising a confusing and/or stressful daily life event that occurred during the past week; 2) formulating a negative and a positive thought based on the chosen event; 3) determining the amount of stress that is evoked by the chosen event; 4) patient focuses on the chosen event while being presented with a distracting stimulus; 5) evaluating the amount of stress that is caused by the chosen event; 6) linking positive thoughts to the negative one when the stress caused by the chosen event does no longer exist; 7) evaluation and closure of session.

SUMMARY:
Rationale: Currently, for youngsters there is no treatment available that directly targets the core symptoms of autism. EMDR is hypothesized to improve the core symptoms of ASD by reducing the generally high stress levels experienced during social interactions, and increasing the functional connectivity in neuronal networks associated with executive functioning and limbic circuitry.

Objective: The primary objective of the study is to determine if EMDR reduces the core symptoms of ASD and daily experienced stress in youngsters diagnosed with ASD.

Study design: Longitudinal multiple single case studies. Study population: Youngsters aged 12-21 years who are diagnosed with ASD and have a full-scale IQ of 80 or more (N=20).

Intervention: 10 weekly EMDR sessions.

Main study parameters/endpoints: The main endpoint of the study are autism symptoms, which will be assessed using the Social Responsiveness Scale (SRS-A) and the Autism Diagnostic Observation Schedule (ADOS 2). The SRS-A will be administered prior, during and after treatment. The ADOS 2 will be administered prior to treatment and after treatment completion. In addition, we will also administer the Trauma Symptom Investigation Form in Autism Spectrum Disorders (TIF-ASD) questionnaire prior to, during, and after treatment. Furthermore, to answer more fundamental questions concerning the working mechanism of EMDR in ASD, other secondary outcome measures (i.e. PSS-10, AWMA-2) will be included.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants are expected to benefit from treatment. The risks associated with study participation are considered negligible and the burden associated with participation is estimated as low.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ASD (with or without comorbid psychiatric disorders, except PTSD and anxiety disorders)
* Full-scale IQ of 80 or more
* Able to understand and speak Dutch

Exclusion Criteria:

* Receiving other treatments than medication on a stable dosage.
* PTSD or other comorbid psychiatric disorders that require immediate and continuous treatment.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in autism symptoms | 0, 1, 2, 3 weeks before intervention; week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 of intervention; 1 and 12 weeks after intervention
  Change in autism symptoms is assessed with the SRS-A, which measures youngsters' ability to engage in reciprocal social behaviour in natural social settings, among all domains of autistic symptoms. The SRS-A consist of 5 subscales: 1) Social Awareness, 2) Social Cognition, 3) Social Communication 4) Social Motivation, and 5) Autistic Mannerisms. In total the five subscales comprise 65-items that are answered on a 4-point scale ranging from never true to almost always true. Completion of the questionnaire takes about 15 minutes. The SRS-A is completed by both parents and youngsters separately. Considering that SRS-A scores provided by youngsters are likely to be less reliable, the total score of the parents will serve as the primary outcome measure. In a secondary analysis, the total score of the youngsters will be used to determine the extent to which they perceive EMDR as an effective treatment.
Change in autism symptoms | 3 weeks before intervention; 1 week after intervention
  Using the Autism Diagnostic Observation Schedule 2 (ADOS 2) changes in autism symptoms prior to and after treatment will be assessed. The ADOS is administered by observing the youngster during a semi-structured observation schedule. With the ADOS, the clinician elicits social, communicative, stereotyped and play behavior to observe symptoms of ASD. Activities are performed with a 40 to 60 minutes protocol. Observations of the clinician are categorized and a score is assigned for each domain of ASD symptoms. Total scores on the ADOS are compared pre-treatment and post-treatment.
Change in autism symptoms | 0, 1, 2, 3 weeks before intervention; week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 of intervention; 1 and 12 weeks after intervention
  Using the Trauma Symptom Investigation Form in Autism Spectrum Disorders (TIF-ASD) changes in autism symptoms prior to, during, and after treatment will be assessed. The TIF-ASD assesses the impact of traumatic events on five core symptoms of autism: 1) social and (verbal) communication skills; 2) behavioral problems; 3) stereotypical & ritualistic behaviors; 4) self-care skills; 5) vegetative symptoms. The total scale consists of 20 items which are completed by an observer (in our case the parents). Items are answered on a 5-point scale ranging from never to always. Completing all items takes about 5 minutes. The TIF-ASD is the only measurement, assessing the traumatic symptoms and behavioral aspects related to ASD due to traumatic events.

SECONDARY OUTCOMES:
Change in disease severity | 3 weeks before intervention; 1 and 12 weeks after intervention
  Youngsters' disease severity and global improvement will be assessed with the Clinical Global Impression Scales (CGI). To assess severity and afterwards improvement, both pre- and post-treatment assessments will be conducted. Assessment are conducted by a clinician who observes a youngster for about 15 minutes while interacting with others. Based on one's past experience with similar patients, the CGI-S enables a clinician to rate the severity of a patient's illness. Severity is assessed on a 7-point scale ranging from not at all ill to extremely ill. Opposed to the CGI-S, the CGI-I enables a clinician to assess the extent to which the severity of a patient's illness has improved or worsened relative to the baseline assessment. Improvement is assessed on a 7-point scale ranging from very much improved to very much worsened.
Change in experienced stress | 0, 1, 2, 3 weeks before intervention; week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10 of intervention; 1 and 12 weeks after intervention
  Experienced stress will be measured by the Perceived Stress Scale-10 (PSS-10) that assess the degree to which individuals find their lives unpredictable, uncontrollable, and overloading. The 10 items are answered on a 5-point scale ranging from never to very often. Completion time is about 3 minutes.
Change in general well-being | 3 weeks before intervention; 1 and 12 weeks after intervention
  General well-being will be measured with the Quality of Life - Questionnaire (QoL-Q). This questionnaire consist of four subscales: satisfaction, competence or productivity, empowerment or independence, and social belonging or community integration, which result in an overall quality of life score. Each subscale contains 10 items, scored on a 3-point scale ranging from not satisfied to very satisfied. Higher scores indicate higher subjective quality of life. Completion time is about 5 minutes.
Change in working memory capacity | 3 weeks before intervention; 1 week after intervention
  Working memory capacity is assessed using the letters mix task of the Alloway Working Memory Assessment (AWMA-2). The task is administered before and after treatment completion. The completion of these task takes about 10 minutes.
Change in working memory capacity | 3 weeks before intervention; 1 week after intervention
  Working memory capacity is assessed using the turning figures task of the Alloway Working Memory Assessment (AWMA-2). The task is administered before and after treatment completion. The completion of these task takes about 10 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Martine Van Dongen-Boomsma, PhD, Principal Investigator — Karakter Child and Adolescent Psychiatry University Centre
Locations (1):
- Karakter kinder- en jeugdpsychiatrie, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No